CLINICAL TRIAL: NCT03377959
Title: Effects of Pilates Method in the Range of Young Ballerina's Turnout
Brief Title: Effects of Pilates Method in the Range of Ballerina's Turnout
Acronym: PilatesTurnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Aline Nogueira Haas, PhD, Federal University of Rio Grande do Sul
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TURN1217
Record Dates: First submitted 2017-12-07; First posted 2017-12-19 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Dancing
Keywords: dance; ballet; Exercise Movement Techniques; turnout

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Group (Experimental): Pilates Method Mat classes and Ballet Classes three times a week, totaling 24 session of each.
  Interventions: Other: Pilates Mat Classes; Other: Ballet Classes
- Ballet Group (Other): Ballet Classes three times a week, totaling 24 sessions.
  Interventions: Other: Ballet Classes

INTERVENTIONS:
Other: Pilates Mat Classes — The intervention, the exercises, and their progressions were systematized based on protocol proposed by Siler (2008).
  Arms: Pilates Group
Other: Ballet Classes — The intervention is ballet classes three times a week, 1 hour and 30 min. The ballet classes consists in barre work and center work with specific ballet exercises.

SUMMARY:
A high degree of turnout is desired by many dancers, because enables an efficient weight transfer; provides an excellent extension and control; and reduces the risk of injury when used properly. The dancer's body conditioning is worked and acquired through various types of training, among which stands out the Pilates Method. Thus, the aim of the study is to determine the effect of a training program of Pilates Method in the range of ballerinas' turnout. The study will be conducted with young dancers, between 10 and 14 years, who practice classical dance twice a week. They will be randomly divided into two groups: intervention and control, but only the intervention group will do Pilates classes. To verify the extent of the turnout, tests will be applied in both groups, before the start of Pilates classes (pre-test) and after 24 sessions (post-test). In the evaluation protocol will be collected kinematic data, while performing the movements of demi plié and elevé. Anthropometric variables of height and body mass will be obtained; and also the extent of the passive and active turnout in dancers.

ELIGIBILITY:
Inclusion Criteria:

* be female; age between 10 and 14 years; have practiced classical ballet classes for at least three years; attend classical ballet classes at least twice a week; have a minimum frequency of 80% during the whole intervention period.

Exclusion Criteria:

* present some injury during intervention period and data collection; have more than two consecutive absences in classical ballet and Pilates classes; not to continue with their routine of physical activities throughout the intervention period.

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
The change in turnout | One week before the first session of the intervention and 12 weeks after the intervention
  Turnout is determined as external rotation of the coxofemoral joint, and is considered perfect when reaching an angle of 180 ° between the longitudinal axis of the feet. The change in turnout will be evaluated one week before the first session of the intervention and after 12 weeks of Mat Pilates training. So, the primary outcome is the change in the range of ballerinas' turnout.

CONTACTS AND LOCATIONS:
Overall Officials: Aline Nogueira Haas, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Laboratório de Pesquisa do Exercício, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Leva P. Adjustments to Zatsiorsky-Seluyanov's segment inertia parameters. J Biomech. 1996 Sep;29(9):1223-30. doi: 10.1016/0021-9290(95)00178-6. PMID 8872282
- [Background] Gilbert CB, Gross MT, Klug KB. Relationship between hip external rotation and turnout angle for the five classical ballet positions. J Orthop Sports Phys Ther. 1998 May;27(5):339-47. doi: 10.2519/jospt.1998.27.5.339. PMID 9580893
- [Background] Koutedakis Y, Sharp NC. Thigh-muscles strength training, dance exercise, dynamometry, and anthropometry in professional ballerinas. J Strength Cond Res. 2004 Nov;18(4):714-8. doi: 10.1519/13983.1. PMID 15574072
- [Background] van Merkensteijn GG, Quin E. Assessment of Compensated Turnout Characteristics and their Relationship to Injuries in University Level Modern Dancers. J Dance Med Sci. 2015 Jun;19(2):57-62. doi: 10.12678/1089-313X.19.2.57. PMID 26045396